CLINICAL TRIAL: NCT02775721
Title: Weight Loss and Gastrostomy Tube Care Outcomes in Head and Neck Cancer Patients With Gastrostomy Tube Placement
Acronym: G-Tube
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: St. John Health System, Oklahoma (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: G-Tube
Record Dates: First submitted 2015-09-23; First posted 2016-05-18 (Estimated); Last update posted 2018-04-17 (Actual); Status verified 2018-04

CONDITIONS: Malnutrition; Gastrostomy
Keywords: Nursing Education; Weight Loss; Gastrostomy Tube Care
MeSH Terms: conditions — Malnutrition; Weight Loss

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Cohort A (Other): Head and Neck Cancer patients receiving Radiation Therapy Only. The purpose is to do a comparative analysis and identify if patient quality of life outcomes are the same, better or worse when compared to Cohorts B and C.
  Interventions: The research nurse will provide gastrostomy tube care education and skin care education at each study visit utilizing the nursing process.
  Speech therapy education and evaluation is assessed per standard of care by the attending speech therapist.
  Nutritional therapy education and evaluation is assessed per the attending dietitian.
  The European Organization for Research and Treatment of Cancer (EORTC) head and neck cancer module (QLQ-H&N35) and EORTC Core Questionnaire (QLQ-C30) version 3.0 will be completed by the subject.
  Interventions: Other: Nursing Education related to Gastrostomy Tube Care; Other: Speech Therapy Education and Evaluation; Other: Nutritional Therapy Education and Evaluation; Other: Quality of Life Questionnaire C30 version 3; Other: Quality of Life Questionnaire EORTC QLO - H&N35
- Cohort B (Other): Head and Neck Cancer patients receiving Chemotherapy Only. The purpose is to do a comparative analysis and identify if patient quality of life outcomes are the same, better or worse when compared to Cohorts A and C.
  Interventions: The research nurse will provide gastrostomy tube care education and skin care education at each study visit utilizing the nursing process.
  Speech therapy education and evaluation is assessed per standard of care by the attending speech therapist.
  Nutritional therapy education and evaluation is assessed per the attending dietitian.
  The European Organization for Research and Treatment of Cancer (EORTC) head and neck cancer module (QLQ-H&N35) and EORTC Core Questionnaire (QLQ-C30) version 3.0 will be completed by the subject.
  Interventions: Other: Nursing Education related to Gastrostomy Tube Care; Other: Speech Therapy Education and Evaluation; Other: Nutritional Therapy Education and Evaluation; Other: Quality of Life Questionnaire C30 version 3; Other: Quality of Life Questionnaire EORTC QLO - H&N35
- Cohort C (Other): Head and Neck Cancer patients receiving Chemotherapy and Radiation therapy. The purpose is to do a comparative analysis and identify if patient quality of life outcomes are the same, better or worse when compared to Cohorts A and B.
  Interventions: The research nurse will provide gastrostomy tube care education and skin care education at each study visit utilizing the nursing process.
  Speech therapy education and evaluation is assessed per standard of care by the attending speech therapist.
  Nutritional therapy education and evaluation is assessed per the attending dietitian.
  The European Organization for Research and Treatment of Cancer (EORTC) head and neck cancer module (QLQ-H&N35) and EORTC Core Questionnaire (QLQ-C30) version 3.0 will be completed by the subject.
  Interventions: Other: Nursing Education related to Gastrostomy Tube Care; Other: Speech Therapy Education and Evaluation; Other: Nutritional Therapy Education and Evaluation; Other: Quality of Life Questionnaire C30 version 3; Other: Quality of Life Questionnaire EORTC QLO - H&N35

INTERVENTIONS:
Other: Nursing Education related to Gastrostomy Tube Care — The research nurse will provide educational intervention at each study visit utilizing the nursing process.
Other: Speech Therapy Education and Evaluation — Speech therapy will be conducted per standard of care, the protocol does not dictate the frequency or treatment plan of care. Speech therapy and evaluation is assessed per the attending speech therapist. The study team will collect all data related to speech therapy education and evaluation at each study visit per protocol. All collected data will be utilized in final protocol analysis.
Other: Nutritional Therapy Education and Evaluation — Nutritional therapy will be conducted per standard of care, the protocol does not dictate the frequency or treatment plan of care. Nutritional therapy and evaluation is assessed per the attending dietitian. The study team will collect all data related to nutritional therapy education and evaluation at each study visit per protocol. All collected data will be utilized in final protocol analysis.
Other: Quality of Life Questionnaire C30 version 3 — 30-item instrument that measures the Health Related Quality of Life (HRQoL) in a wide range of cancer patient populations.
Other: Quality of Life Questionnaire EORTC QLO - H&N35 — 35-item instrument that measures the Health Related Quality of Life specific to Head and Neck cancer patient populations.

SUMMARY:
Poor nutritional status and malnutrition are prevalent for patients undergoing treatment for head and neck cancer. Inadequate dietary intake is multi factorial, with patients experiencing dysphagia and or anorexia caused by various cancer treatments. Current standard practice utilizes Gastrostomy Tube placement to manage adverse nutritional effects related to Head and Neck cancer treatment.

DETAILED DESCRIPTION:
The purpose of this study is to assess the quality of life and educational intervention outcomes of Head and Neck Cancer patients who have a gastrostomy tube placed per standard of care.

A high incident of Gastrostomy tube replacement occurs related to clogged, dislodged, and/or pulled out tubes. In addition, patients not eating or drinking after Gastrostomy tube placement, compounded by complications related to radiation treatment, results in decreased swallowing function. Inadequate swallow function, especially when combined with inadequate use of Gastrostomy tube, due to non-functional tube or insufficient patient knowledge in use of tube, results in poor nutritional status and excessive weight loss.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older
* Head and Neck cancer diagnosis
* Esophageal cancer diagnosis
* Receiving chemotherapy and/or radiation therapy
* Gastrostomy Tube placed within the last 30days or scheduled to have a gastrostomy tube placed within the next 30 days

Exclusion Criteria:

* Not eligible for chemotherapy and/or radiation therapy
* Unwilling or unable to sign informed consent
* Any cognitive or mental deficits that would prevent patient from completing questionnaires or understanding educational interventions
* Current pre-existing Gastrostomy tube complications if a current Gastrostomy tube is in place prior to informed consent (i.e., skin breakdown, tube breakdown, other tube complications).
* No Gastrostomy tube placement
* Non-English Speaking

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2015-07; Primary Completion 2018-12 (Estimated); Study Completion 2018-12 (Estimated)

PRIMARY OUTCOMES:
Sustained ± 10% body weight post gastrostomy tube placement for cancer therapy treatment. | through study completion, an average of 2 years
  Patient Reported Outcomes utilizing EORTC QLQ-C30 version 3 and EORTC QLO - H&N35 Questionnaires.
Patient loss of speech increase or decrease | through study completion, an average of 2 years
  Measure functional status of speech therapy every 30 days
Patient loss of swallow function increase or decrease | through study completion, an average of 2 years
  EORTC QLO - H&N35 Questionnaire

SECONDARY OUTCOMES:
Patient knowledge of management and care of Gastrostomy Tube. | through study completion, an average of 2 years
  Nursing Education utilizing the Gastrostomy Tube education booklet will improve patient's knowledge and management of Gastrostomy Tube care
Maintaining swallowing function | through study completion, an average of 2 years
  Speech therapy
Patient Reported Outcomes utilizing EORTC QLQ-C30 version 3 Questionnaire. | through study completion, an average of 2 years
  Assess Quality of Life
Patient Reported Outcomes utilizing EORTC QLO - H&N35 Questionnaire. | through study completion, an average of 2 years
  Assess Quality of Life

CONTACTS AND LOCATIONS:
Overall Officials: Candida Barlow, MSN RN, Principal Investigator — St. John Health System
Locations (1):
- St. John Health System, Tulsa, Oklahoma, United States

IPD SHARING:
Plan to Share IPD: Undecided